CLINICAL TRIAL: NCT03676387
Title: Prediction of Optimal Pediatric Endotracheal Tube Size "Aged Based Formula Versus Ultrasonography"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nevert Adel, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MansouraU1
Record Dates: First submitted 2018-09-11; First posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Anesthesia Intubation Complication
Keywords: pediatric; endotracheal tube; ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aged based group (group AB) (n = 27) (No Intervention): ETT size was determined according to age
- Ultrasound based group (group UB) (n = 27): ETT was determined (Active Comparator): ETT was determined according to the subglottic transverse diameter that was estimated with ultrasonography.
  Interventions: Other: ultrasound guided

INTERVENTIONS:
Other: ultrasound guided — Ultrasonography technique:
  The subglottic diameter was estimated with B-mode ultrasonography (Korean, Siemens, Acuson, x300) with a 10-13-MHz linear probe positioned on the midline of the anterior neck (figure1). The evaluation began by identifying the true vocal folds as paired hyperechoic linear structures that moved with respiration and swallowing before patients were paralyzed. The probe was then moved caudally to visualize the cricoid arch which appears as an arched, rounded and hypoechoic structure (figure2). The transverse air-column diameter was measured at the lower edge of the cricoid cartilage after patients were paralyzed (figure3).
  The measurements of the subglottic diameter was used to select the outer diameter of endotracheal tube by the equation [ETT OD=0.55*(subglottic diameter)+1.16] (Shibasaki et al., 2010), since the outer diameter of endotracheal tube differs among different manufactures, we used uncuffed Mallinckrodt tracheal tube with a Murphy's eyes.
  Arms: Ultrasound based group (group UB) (n = 27): ETT was determined

SUMMARY:
Background: Ultrasound (US) imaging technique has recently emerged as a novel, simple, portable, noninvasive tool helpful for airway assessment and management. Initial few published reports were on soft tissue imaging of neck, focusing on pre-tracheal structure and anterior tracheal wall. In our study, we compared the measurement of subglottic diameter using ultrasonography and the aged based formula in prediction of endotracheal tube size in children underwent elective surgical operation under general anesthesia.

Methods: Patients were randomly divided in 2 groups (27 patients each) using a computer-generated randomization schedule. The first group was aged based group (group AB) (n = 27): the endotracheal tube size was determined according to age of the child [inner diameter [ID] in mm = (age in yr/4) +4. The second group was ultrasound based group (group UB) (n = 27): the endotracheal tube size was determined according to the subglottic transverse diameter that was estimated with ultrasonography (the outer diameter of endotracheal tube (ETT OD) = 0.55*(subglottic diameter)+1.16) .

DETAILED DESCRIPTION:
Introduction:

Pediatric tracheal intubation requires considerable expertise and can represent a challenge to many anesthesiologists(Marciniak et al.,2009). Anatomically; the larynx of a pediatric patient assumes a funnel shape with its narrowest part at the level of the cricoid ring, which cannot be seen during conventional laryngoscopy (Karsli et al.,2002).

Choosing the correct endotracheal tube (ETT) size needed for intubation of pediatric patients is important because an inappropriately too large tracheal tube can cause upper airway damage (e.g., local ischemia, ulceration, scar formation) and the potential for subsequent subglottic stenosis. In contrast, an ETT that is too small may result in insufficient ventilation, poor reliability of end-tidal gas monitoring, leakage of anesthetic gases into the operating room environment, and an enhanced risk of aspiration(Karsli et al.,2002).

Different algorithms and formula have been proposed to choose the best-fitting size of the endotracheal tube. Age-based formulas, such as those of Cole and Motoyama, have been used to estimate optimal ETT size for more than half a century (Motoyama,1990) and this formula is [inner diameter (ID) in mm = (age in yr/4) +4]. Predictive formulas for appropriate ETT size have also been based on patient weight and height as[ID in mm = 2 + height in cm/30] and [ID in mm = 2.44 + age in yr ×0.1 + height in cm ×0.02 + weight in kg ×0.016] and other formula as the width of the 5th fingernail is used for ID prediction of the ETT [ID in mm = maximum width of the 5th fingernail] (Shibasaki et al.,2010). However, these methods are not always suitable because the size of the airway varies considerably between patients.

Ultrasound guided is helpful for evaluate the subglottic transverse diameter which is safe , sample, painless and non invasive modality for prediction of proper endotracheal tube size (Jagadish G Sutagatti et al., 2017).

In this study, we compared the measurement of subglottic diameter using ultrasonography and the aged based formula in prediction of endotracheal tube size in children underwent elective surgical operation under general anesthesia.

Patients and methods:

Study design and participants After getting approval from the institutional research board(MS/16.01.143), faculty of medicine , Mansoura University, written informed consents were obtained from parents of fifty children aged from 1 to 6 years of either sex scheduled for elective surgery not exceeded 90 minutes underwent general anesthesia with uncuffed endotracheal tube. This randomized controlled study was conducted in Emergency Hospital, Mansoura University between April/2016 to April/2017 .

Patient exclusion criteria include: an anticipated difficult airway, any respiratory disease that might cause airway narrowing, pre-exiting laryngeal or tracheal pathology, any lesion that could cause airway deformity due to fibrosis or the presence of a neck anatomical pathologies that might have unpredictable effect on the ultrasound assessment of the airway and prolonged surgery more than 90 minutes .

Sample size calculation:

The appropriateness of ETT size was adopted as a primary parameter for effective size used for sample size calculation. A power of 80% was accepted with alpha error of 0.05. fifty four patients in both groups were found to be enough to detect a 20% difference between groups.

Patients were randomly divided in 2 groups (27 patients each) using a computer-generated randomization schedule.

Aged based group (group AB) (n = 27): ETT size was determined according to age of the child, inner diameter [ID] in mm = (age in yr/4) +4(Van den Berg and Mphanza, 1997).

Ultrasound based group (group UB) (n = 27): ETT was determined according to the subglottic transverse diameter that was estimated with ultrasonography.

Technique:

On arrival to the operating room, basic monitors were applied {ECG, pulse oximetry, non-invasive blood pressure (NIBP)}, baseline values were recorded and An intravenous cannula (24G) was inserted and secured . General anesthesia was induced by inhalation of sevoflurane. Muscular relaxation was achieved with atracurium (0.5mg/kg) to facilitate the endotracheal intubation under direct laryngoscopy. The patients were ventilated with sevoflurane in 100% oxygen via a facemask before intubation for 3 min for proper muscles relaxation. ETT was chosen according to each group. Aged based formula (inner diameter [ID] in mm = (age in yr/4) +4) was used in group AB and in group UB, during mask ventilation ultrasound guided subglottic transverse diameter was measured with assistant anesthesiologist help. To avoid observer bias by anesthesiologist who performs the leak test by the absence of ultrasound machine in the operating room, the ultrasound assessment also was done in group AB(aged-based).

Ultrasonography technique:

The subglottic diameter was estimated with B-mode ultrasonography (Korean, Siemens, Acuson, x300) with a 10-13-MHz linear probe positioned on the midline of the anterior neck (figure1). The evaluation began by identifying the true vocal folds as paired hyperechoic linear structures that moved with respiration and swallowing before patients were paralyzed. The probe was then moved caudally to visualize the cricoid arch which appears as an arched, rounded and hypoechoic structure (figure2). The transverse air-column diameter was measured at the lower edge of the cricoid cartilage after patients were paralyzed (figure3).

The measurements of the subglottic diameter was used to select the outer diameter of endotracheal tube by the equation [ETT OD=0.55*(subglottic diameter)+1.16] (Shibasaki et al., 2010), since the outer diameter of endotracheal tube differs among different manufactures, we used uncuffed Mallinckrodt tracheal tube with a Murphy's eyes.

The inner diameter of endotracheal tube that was calculated according to table (1) which show the correlation between outer and inner diameter of the endotracheal tube.

Determination of appropriateness of ETT size:

Another anesthesiologist who was blinded to the group allocation did the air leak test in all patients. The air leak test was done after successful intubation of ETT chosen on the basis of either of two methods, The correct tracheal tube size was considered optimal when an audible air leak around the tube at an inspiratory airway pressure was detected between 10-30 cm H2O, with the head and neck in a neutral position. The presence of an air leak was assessed by closing off the pop-off valve and allowing pressure to rise slowly until an audible leak was heard using a stethoscope on the tube. If there was no audible leak when the lung were inflated to a pressure of 30 cm H2O, the tube was exchanged with one that was 0.5 mm smaller. But if a leak occurred at an inflation pressure of less than 10 cm of H2O, the ETT was exchanged for one with the 0.5 mm larger tube.

The following parameters were monitored:

1. Primary outcome: Number of optimum tube selection was monitored in both group (group AB and group UB).2- Number of reintubation due to large or small tube.
2. Secondary outcome: 1- Time of intubation. 2- Complication after extubation.

Statistical analysis:

All statistical analyses were performed using SPSS for windows version 20.0 (SPSS, Chicago, IL). Continuous data we re-expressed in mean ±standard deviation (SD) white categorical data were expressed in number and percentage. The differences between two groups were determined using Student's t test for variables with continuous data and chi-square test for variables with categorical data. The 95% confidence interval (CI) for the frequency of correct size of the endotracheal tube (ETT) was calculated. Statistical significance was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* fifty four children aged from 1 to 6 years of either sex
* scheduled for elective surgery not exceeded 90 minutes
* underwent general anesthesia with uncuffed endotracheal tube.

Exclusion Criteria:

* an anticipated difficult airway
* any respiratory disease that might cause airway narrowing
* pre-exiting laryngeal or tracheal pathology
* any lesion that could cause airway deformity due to fibrosis or the presence of a neck anatomical pathologies that might have unpredictable effect on the ultrasound assessment of the airway
* prolonged surgery more than 90 minutes .

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-04-16 (Actual); Study Completion 2017-04-16 (Actual)

PRIMARY OUTCOMES:
1- Number of optimum tube selection was monitored in both group (group AB and group UB) (number and percentage %). | 1 year
Number of reintubation due to large or small tube (number and percentage %). | 1 year

SECONDARY OUTCOMES:
Time of intubation (minutes). | 1 year
complication after extubation | 1 year